CLINICAL TRIAL: NCT03005899
Title: Double-Blind, Placebo-Controlled Comparative Study of SyB P-1501 (Fentanyl HCI) for Treatment of Postoperative Pain
Brief Title: Study of SyB P-1501 (Fentanyl HCI) for Treatment of Postoperative Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Clinical trial was terminated due to discontinuation of drug product by the investigational drug supplier.
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015002
Record Dates: First submitted 2016-11-10; First posted 2016-12-30 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- SyB P-1501 group (Experimental): One patch of SyB P-1501 contains 10.8 mg of fentanyl hydrochloride (fentanyl 9.7 mg) and produces an electric current to deliver the drug iontophoretically after the system is activated. 40 µg fentanyl per on-demand dose, each delivered over 10 minutes for a maximum of 6 doses/hr for 24 hours or maximum of 80 doses. Each system will inactivate at 80 doses or 24 hours, whichever occurs first.
  Interventions: Drug: SyB P-1501
- SyB P-1501 placebo group (Placebo Comparator): Identical to SyB P-1501 containing hydrogel that contains the active ingredient fentanyl HCI in its structure and appearance but production of an electric current and subsequent drug administration by iontophoresis are prevented because of its modified circuit.
  Interventions: Drug: SyB P-1501 placebo

INTERVENTIONS:
Drug: SyB P-1501 — After extubation and adequate titration by Fentanyl intravenous injection, the investigational product is applied to outer upper arm or chest on patient who confirmed treatment eligibility. Fentanyl 40 μg per dose is delivered over a 10-minute period by pressing the dosing button by the subject as needed. The 10-minute dosing period is a system lock-out time, allowing for a maximum of 6 doses per hour. One system is operable for 24 hours or until 80 doses are delivered, whichever occurs first.
  Duration of application of the investigational product is 24 hours. Duration of application may be extended for up to 72 hours or until the third system is used, whichever occurs first, if the patient requests it and the specified tests can be performed
  Arms: SyB P-1501 group
Drug: SyB P-1501 placebo — Identical to SyB P-1501 containing hydrogel that contains the active ingredient fentanyl HCI in its structure and appearance but production of an electric current and subsequent drug administration by iontophoresis are prevented because of its modified circuit.
  Arms: SyB P-1501 placebo group

SUMMARY:
This is a Phase 3 clinical trial to compare the safety and efficacy of SyB P-1501 with the SyB P-1501 placebo for the management of the first 24 hours of post-operative pain.

ELIGIBILITY:
Patients who meet all of the inclusion criteria from the day of informed consent to one day before surgery and to whom none of the exclusion criteria is applicable will be eligible to participate in the study.

Inclusion Criteria:

1. Expected to require opioid analgesia for management of post-operative pain for at least 24 hours after surgery and require postoperative pain control
2. Underwent one of the following surgeries under general anesthesia:

   * Abdominal surgery (e.g., gastrointestinal, gynecological)
   * Orthopedic surgery (e.g., spinal surgery)
   * Thoracic surgery (e.g., respiratory surgery not requiring chest tubes after surgery)
3. ASA physical status I, II or III
4. Age: At least 20 years
5. Sex: Men or women (negative pregnancy test for women of childbearing potential).
6. Inpatient/outpatient status: Inpatient
7. Received adequate information about the study and gave a written consent to participate in the study by himself/herself

Exclusion Criteria:

1. Expected to use continuous intra-operative and post-operative analgesia with local pain control techniques (e.g., spinal/epidural analgesia, nerve block)
2. Scheduled for body surface surgery (e.g., burn, breast reconstruction, skin grafting)
3. Hypersensitive/allergic to fentanyl, skin adhesive and/or cetylpyridinium chloride
4. Expected/scheduled to undergo additional surgical procedure within 36 hours post-operation
5. Known or suspected opioid tolerance
6. Skin disorder that precludes application of investigational product
7. Increased intracranial pressure
8. Concomitant asthma, severe respiratory disorder
9. Having had convulsive seizure attacks within 5 years
10. Patient with medical devices implanted in the body, such as cardiac pacemakers or implantable defibrillators
11. History of opioid, drug and/or alcohol abuse
12. Women who are pregnant, might be pregnant, or are breastfeeding
13. Using any investigational drug, used any investigational drug within the last 6 months
14. Otherwise determined ineligible to participate in the study at the discretion of the principal investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of dropouts due to inadequate analgesia judged by patients or investigator during the period between Hour 3 and Hour 24 of system application | 3 to 24 hours
  proportion of dropouts due to inadequate analgesia during the period between Hour 3 and Hour 24 of system application. Inadequate analgesia cases are defined below.
  * The subject wishes to discontinue the study due to inadequate analgesia
  * Investigator or sub-investigator judges that the patient is to be discontinued due to inadequate analgesia
  * The subject who completes 80 doses within 24 hours is not willing to use the second system and wishes an alternative analgesia

SECONDARY OUTCOMES:
Proportion of dropouts due to inadequate analgesia judged by patients or investigator during the period between the start and Hour 24 of system application | 0 to 24 hours
  Proportion of dropouts due to inadequate analgesia during the period between the start and Hour 24 of system application. Inadequate analgesia cases are defined below.
  * The subject wishes to discontinue the study due to inadequate analgesia
  * Investigator or sub-investigator judges that the patient is to be discontinued due to inadequate analgesia
  * The subject who completes 80 doses within 24 hours is not willing to use the second system and wishes an alternative analgesia
time to dropout during the period between Hour 3 and Hour 24 of system application (Non-dropout: censored at 24 hours after application) or from application (Non-dropout: censored at 24 hours after application) | 0 to 24 hours
  Time to dropout during the period between Hour 3 and Hour 24 of system application will be evaluated (Non-dropout: censored at 24 hours after application).
  Time to dropout from application will be also evaluated (Non-dropout: censored at 24 hours after application)
Proportion of dropouts for any reason during the period between Hour 3 and Hour 24 of system application or between the system application and Hour 24 | 0 to 24 hours
  Proportion of dropouts for any reason during the period between Hour 3 and Hour 24 of system application will be evaluated.
  Proportion of dropouts for any reason between the system application and Hour 24 will be also evaluated.
pain intensity（Numerical rating scale: NRS） expressed as a mean for each group and compared using Student t test between groups | 0 to 72 hours
  During the pre-treatment period, up to Hour 24 of the treatment period, and at the time of removing each patch, pain intensity at the time of each measurement will be evaluated as NRS
Patient global assessment of method of Pain Control compared using Wilcoxon two sample test or Fisher's exact test between groups | 0 to 24 hours
  Patient global assessment of therapeutic effect at the end of Hour 24 or when the study treatment is discontinued will be evaluated on a categorical scale
Investigator global assessment of method of Pain Control compared using Wilcoxon two sample test or Fisher's exact test between groups | 0 to 24 hours
  Investigator global assessment of therapeutic effect at the end of Hour 24 or when the study treatment is discontinued will be evaluated on a categorical scale
Adverse events (including application site erythema and other application site reactions) coded with MedDRA and graded for severity at three level | 20 days
  Adverse event evaluation (including application site erythema and other application site reaction)
Changes in the measurements of vital signs (blood pressure, heart rate, respiratory function, SpO2) and laboratory tests (hematological test and blood biochemical test) measured with descriptive statistics | 20 days
  Changes in the measurements of vital signs (blood pressure, heart rate, respiratory function, SpO2) and laboratory tests (hematological test and blood biochemical test)
incidence of technical failures defined as unfavorable conditions concerned with such as quality, safety, or performance of mechanic parts of investigational products | 20 days
  Presence or absence and evaluation of technical failures

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Kawashima, Study Director — SymBio Pharmaceuticals
Locations (29):
- Japan (29):
  - Research Site, Nagakute, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyoake, Aichi-ken
  - Research Site, Kobe, Hyōgo
  - Research Site, Kahoku, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Hiragi, Kagawa-ken
  - Research Site, Nankoku, Kochi
  - Research Site, Sendai, Miyagi
  - Research Site, Matsumoto, Nagano
  - Research Site, Kashihara, Nara
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Sayama, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Takatsuki, Osaka
  - Research Site, Izumo, Shimane
  - Research Site, Arakawa City, Tokyo
  - Research Site, Minato, Tokyo
  - Research Site, Yonago, Tottori
  - Research Site, Ube, Yamaguchi
  - Research Site, Chūō, Yamanashi
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Kagoshima
  - Research Site, Kyoto
  - Research Site, Okayama
  - Research Site, Saga
  - Research Site, Tokushima
  - Research Site, Wakayama